CLINICAL TRIAL: NCT07060118
Title: Gluten Free Diet For Treatment of Symptoms of Hashimoto's Hypothyroidism
Brief Title: Gluten Free Diet in Hashimoto's Hypothyroidism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Keren Zhou, Research Director, The Cleveland Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 25-472
Record Dates: First submitted 2025-06-23; First posted 2025-07-11 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Hypothyroidism; Hashimoto Disease
MeSH Terms: conditions — Hypothyroidism; Hashimoto Disease | interventions — Diet, Gluten-Free

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gluten Free Diet in Hashimoto's Hypothyroidism (Experimental)
  Interventions: Dietary Supplement: Gluten Free Diet in Hashimoto's Hypothyroidism

INTERVENTIONS:
Dietary Supplement: Gluten Free Diet in Hashimoto's Hypothyroidism — Gluten Free Diet in patients with Hashimoto's Hypothyroidism

SUMMARY:
Hashimoto's thyroiditis is an autoimmune condition that reduces functioning of the thyroid gland and can lead to a substantial decline in quality of life for patients, with impacted patients often describing unremitting brain fog, fatigue/malaise and weight gain leading to difficulty functioning in their jobs and homes. It is the most common cause of hypothyroidism in the U.S. and affects up to 10% of the global population. The typical treatment for Hashimoto's is thyroid hormone replacement with medications such as levothyroxine. However, despite adequate treatment as defined by thyroid hormone levels within the reference range, up to 10% of patients will experience persisting symptoms which can dramatically impair quality of life. While various theories have been postulated for the residual symptoms, several studies indicate that they are related to the thyroid autoimmunity, specifically the autoantibodies that are made by the immune system in Hashimoto's thyroiditis in response to the thyroid (ie thyroid peroxidase [TPO], thyroglobulin [Tg] antibody [AB]) and the associated inflammation with the immune response. Removal of thyroid (ie total thyroidectomy) reduces levels of these thyroid antibodies and results in significant improvement in quality-of-life. However, thyroidectomy is an invasive procedure with potential for morbidity such as damage to the recurrent laryngeal (nerve that controls the vocal cords and thus speech), bleeding and infection, so there is interest in other more conservative modalities for lowering the inflammation and autoimmune burden in Hashimoto's thyroiditis.

In an effort to identify a less invasive approach for reducing the levels of thyroid antibodies and inflammation, attention has moved to the intersection of Hashimoto's thyroiditis and the gut. Hashimoto's has a strong association with autoimmune disorders impacting the gastrointestinal tract, in particular celiac disease and non-celiac gluten sensitivity (NCGS). NCGS is a condition where there are intestinal and extra-intestinal symptoms associated the consumption of gluten but no presence of anti-tissue transglutaminase antibodies (anti-tTG) which define Celiac Disease. This connection between Hashimoto's thyroiditis and sensitivity to gluten appears to be not only genetic, as those with Celiac Disease/NCGS and Hashimoto's thyroiditis have common HLA haplotypes, but also at the level of the intestine with gut microbiome dysfunction.

DETAILED DESCRIPTION:
Researchers postulate increased intestinal permeability in those with NCGS exposed to gluten leading to immune activation and propagation of autoimmunity on the thyroid. Hence, elimination of gluten in diet may improve the autoimmunity and inflammation association with Hashimoto's thyroiditis, leading to improvement in negative symptoms such as the fatigue and brain fog.

ELIGIBILITY:
Inclusion Criteria

1. Diagnosis of Hashimoto's thyroiditis
2. Self-perception of reduced quality of life since diagnosis as determined by a ThyPRO score greater than or equal to 35 (higher score suggests lower quality-of-life) based on prior studies reporting of average score in individuals with symptomatic hypothyroidism.
3. Hypothyroidism requiring use of thyroid hormone replacement >6 months prior initiation of study
4. Thyroid hormone levels (TSH, Free T4 and Free T3 as available) within the normal reference range within 3 months of the study initiation
5. Anti-TPO AB greater than or equal to 500 IU/mL and/or Anti-Tg AB greater than or equal to 50 IU/mL at any point in medical history

Exclusion Criteria

1. Prior surgical intervention on thyroid
2. Prior Celiac Disease diagnosis or symptoms which are highly suggestive of undiagnosed Celiac Disease (i.e. chronic diarrhea, blood in stool, unintentional weight loss, family history, etc). In the case of the latter, patients will be directed to speak with their physician to consider screening before being considered for enrollment into the study.
3. Pregnancy
4. Use of gluten-free diet within prior 6 months
5. Active malignancy undergoing treatment
6. Any condition which, based on the investigator's medical judgment, would preclude patient ability to complete the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Primary outcome | 6 months
  Change in quality-of-life metrics

OTHER OUTCOMES:
Outcome measure #2 | 6 months
  Change in thyroid autoantibody titers and hormone levels
Outcome measure #3 | 6 months
  Adherence to gluten free diet
Outcome measure #4 | 6 months
  Correlation of baseline in wheat/gluten proteome reactivity and autoimmunity levels with response to a gluten free diet in terms of thyroid indices and quality-of-life metrics.

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No